CLINICAL TRIAL: NCT02345265
Title: A Phase 2 Study of Olaparib and Cediranib for the Treatment of Recurrent Ovarian Cancer
Brief Title: Testing the Combination of the Study Drugs Cediranib and Olaparib in Recurrent Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00051; NCI-2015-00051 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-700; 9825 (Other: Dana-Farber - Harvard Cancer Center LAO); 9825 (Other: CTEP); UM1CA186644 (NIH); UM1CA186686 (NIH); UM1CA186690 (NIH); UM1CA186691 (NIH); UM1CA186704 (NIH); UM1CA186709 (NIH); UM1CA186712 (NIH); UM1CA186716 (NIH); UM1CA186717 (NIH); ZIABC011078 (NIH)
Record Dates: First submitted 2015-01-23; First posted 2015-01-26 (Estimated); Results first posted 2023-03-28 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-07

CONDITIONS: Fallopian Tube Carcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Ovarian Carcinoma; Ovarian High Grade Endometrioid Adenocarcinoma; Ovarian High Grade Serous Adenocarcinoma; Primary Peritoneal Carcinoma; Primary Peritoneal Endometrioid Adenocarcinoma; Primary Peritoneal Serous Adenocarcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Biopsy; Specimen Handling; cediranib; Magnetic Resonance Spectroscopy; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (olaparib and cediranib maleate) (Experimental): Patients receive olaparib PO BID and cediranib maleate PO QD on days 1-28. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo a biopsy of tumor, blood sample collection, MUGA or echocardiogram, and CT scan or MRI scan throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cediranib Maleate; Procedure: Computed Tomography; Procedure: Echocardiography Test; Procedure: Magnetic Resonance Imaging; Procedure: Multigated Acquisition Scan; Drug: Olaparib; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy of tumor
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cediranib Maleate — Given PO
  Other Names: AZD2171; AZD2171 Maleate; Recentin
Procedure: Computed Tomography — Undergo CT scan
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo echocardiogram
  Other Names: EC; Echocardiography
Procedure: Magnetic Resonance Imaging — Undergo MRI scan
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies how well olaparib and cediranib maleate work in treating patients with ovarian, primary peritoneal, or fallopian tube cancer that has come back after a period of improvement (recurrent). Olaparib and cediranib maleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the association of BROCA-homologous recombination (HR) with the clinical activity of cediranib maleate (cediranib)/olaparib, as measured by progression-free survival (PFS), in women with recurrent platinum-sensitive ovarian cancer.

II. To assess the clinical activity of cediranib/olaparib, as measured by objective response, in women with recurrent platinum-resistant ovarian cancer.

SECONDARY OBJECTIVES:

I. To assess overall survival (OS), objective response, and clinical benefit (stable disease [SD] or response >= 16 weeks) in women with platinum-sensitive ovarian cancer, and PFS, OS, and clinical benefit in women with platinum-resistant ovarian cancer.

II. To assess the safety of cediranib/olaparib in women with recurrent platinum-sensitive and -resistant ovarian cancer.

III. To evaluate the association of circulating endothelial cells at baseline and day 3 with the clinical activity of cediranib/olaparib, as measured by PFS, in women with platinum-sensitive and -resistant ovarian cancer.

IV. To evaluate changes in BROCA-HR status between archival and pre-treatment biopsy samples.

V. To evaluate the associate of BROCA-HR with the clinical activity of cediranib/olaparib as measured by PFS, in women with platinum-resistant ovarian cancer.

VI. To characterize genomic alteration by whole exome sequencing in women with platinum-sensitive and -resistant ovarian cancer.

VII. To identify biomarker signatures that correlate with the clinical activity of cediranib/olaparib in women with recurrent platinum-sensitive and -resistant ovarian cancer, including changes in gene expression or acquired mutations in on-treatment tumor biopsies that are associated with clinical activity, and changes in gene expression or acquired mutations in post-progression biopsies that are associated with clinical resistance.

VIII. To explore changes in biomarker signatures and candidate angiogenic markers from pre-treatment to post-progression in women with platinum-sensitive and -resistant ovarian cancer.

IX. To evaluate the population pharmacokinetics (PK) of the combination of cediranib and olaparib (tablets) in platinum-sensitive and -resistant ovarian cancer.

EXPLORATORY OBJECTIVES:

I. To determine the feasibility of a mobile phone application (app) ecediranib-olaparib (eCO) to collect patient-generated blood pressure and symptom data based upon study protocol recommendations.

II. Assess patient and health care professional perceived usability and satisfaction of the eCO app (for patients) and of a connected web portal (for health care providers).

III. Assess the number of generated alerts to the study team (via the web portal and email "high" alerts) based on pre-determined severity levels.

OUTLINE:

Patients receive olaparib orally (PO) twice daily (BID) and cediranib maleate PO once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo a biopsy of tumor, blood sample collection, multigated acquisition scan (MUGA) or echocardiogram, and computed tomography (CT) scan or magnetic resonance imaging (MRI) scan throughout the study.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed ovarian cancer, peritoneal cancer or fallopian tube cancer and must have a histological diagnosis of either high grade serous or high grade endometrioid cancer based on local histopathological findings; participants with a deleterious BRCA-mutation on a commercial Clinical Laboratory Improvement Amendments (CLIA) assay with other high-grade histologies are also eligible

  * Due to the long acceptance of BRCA testing through Myriad, Myriad testing will be accepted as documentation of a deleterious mutation; if testing for BRCA is done by other organizations, documentation from a qualified medical professional (e.g., ovarian cancer specialty physician involved in the field, high risk genetics physician, genetics counselor) listing the mutation and confirming that the laboratory results show a recognized germline deleterious BRCA1 or BRCA2 mutation or BRCA rearrangements is required to document the presence of a deleterious mutation
* Participants must have measurable disease via Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan, MRI, or calipers by clinical exam
* Patients may not have received prior poly ADP ribose polymerase (PARP) inhibitors
* Patients may have received but may not have progressed on prior anti-angiogenic therapy in the upfront setting
* For platinum sensitive cohort

  * Cancer that has not progressed within 6 months of the last receipt of platinum-based chemotherapy
  * No limit on the number of platinum-based lines
  * No more than one prior non-platinum based line of therapy in the recurrent setting
* For platinum-resistant or -refractory cohort

  * Disease that has progressed within 6 months of the last receipt of platinum-based chemotherapy
  * No more than 1 prior line of therapy in the platinum-resistant/-refractory setting
  * No limit on number of prior lines received in the platinum-sensitive setting prior to development of platinum-resistance (defined as disease progression within 6 months of platinum-based chemotherapy)
* Hormonal therapies used as single agents (i.e. tamoxifen, aromatase inhibitors) will not count towards line limit considerations
* Age >= 18 years of age. Because no dosing or adverse event data are currently available on the use of cediranib or olaparib in patients under the age of 18, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 10 g/dL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x the institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional upper limit of normal
* Creatinine less than or equal to the institutional upper limit of normal or creatinine clearance >= 60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal
* Proteinuria less than or equal to 1+ proteinuria on two consecutive dipsticks taken no less than week apart, or a urine protein:creatinine (UPC) ratio of =< 1
* Coagulation parameters (international normalized ratio [INR], activated partial thromboplastin time [aPTT]) =< 1.25 x ULN institutional limits, except where a lupus anti-coagulant has been confirmed
* Presence of biopsiable disease and willingness to undergo pre-treatment and on-treatment biopsy
* The effects of olaparib and cediranib on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and up to 3 months after end of treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Adequately controlled thyroid function, with no symptoms of thyroid dysfunction and thyroid stimulating hormone (TSH) less than or equal to the upper limit of normal
* Patients must be able to tolerate oral medications and not have gastrointestinal illnesses that would preclude absorption of cediranib or olaparib
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to release and confirmed availability of archival tissue sample for research purposes
* Willingness and ability to check and record daily blood pressure readings; blood pressure cuffs will be provided to patients

Exclusion Criteria:

* Participants may not have had chemotherapy or radiation therapy (RT) within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study and must have recovered to =< grade 1 from adverse events due to agents administered more than 3 weeks earlier; patients should not have received hormonal therapy for treatment of their cancer within 2 weeks of study entry
* Participants should not have received any other investigational agents nor have participated in an investigational trial within the past 4 weeks
* Participants may not have had prior use of PARP inhibitors; patients may not have received prior treatment affecting the VEGF pathway in the recurrent setting, including but not limited to thalidomide, bevacizumab, sunitinib, or sorafenib
* Participants may not have any evidence of ongoing inadequately controlled hypertension (defined as a systolic blood pressure [BP] of > 140 mmHg or a diastolic BP of > 90 mmHg); patients with hypertension may not be on more than three antihypertensive medications for management of their blood pressure (medications that combine two anti-hypertensives into one are considered as two medications); it is strongly recommended that patients who require three antihypertensive medications for baseline management of pre-existing hypertension be actively followed by a cardiologist or blood pressure specialist for management of BP while on protocol
* Participants may not have had any prior history of hypertensive crisis or hypertensive encephalopathy
* Participants may not have had history of abdominal fistula or gastrointestinal perforation; patients with a history of abdominal fistula will be considered eligible if the fistula has healed or was surgically repaired, there has been no evidence of fistula for at least 6 months, and patient is deemed to be at low risk of recurrent fistula
* Participants may not have had a history of intra-abdominal abscess within the past 3 months
* Participants may not have current signs and/or symptoms of bowel obstruction or signs and/or symptoms of bowel obstruction within 3 months prior to starting study drugs
* Participants may not have a dependency on intravenous (IV) hydration or total parenteral nutrition (TPN)
* Participants with any concomitant or prior invasive malignancies are ineligible with the following exceptions:

  * Treated limited-stage basal cell or squamous cell carcinoma of the skin
  * Carcinoma in situ of the breast or cervix
  * Primary endometrial cancer meeting the following conditions: stage not greater than IA, grade 1 or 2, no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell, or other International Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions
  * Prior cancer treated with curative intent with no evidence of recurrent disease 3 years following diagnosis and judged by the investigator to be at low risk of recurrence
* Participants with any of the following:

  * History of myocardial infarction within six months
  * Unstable angina
  * New York Heart Association (NYHA) classification of III or IV
* If cardiac function assessment is clinically indicated or performed: participants will be ineligible if left ventricular ejection fraction (LVEF) is less than normal per institutional guidelines, or < 55%, if the threshold for normal is not otherwise specified by institutional guidelines
* Patients with any of the following risk factors should have a baseline cardiac function assessment:

  * Prior treatment with anthracyclines
  * Prior treatment with trastuzumab
  * Prior central thoracic radiation therapy (RT), including RT to the heart
  * History of myocardial infarction within 6 to 12 months (patients with history of myocardial infarction within 6 months are excluded from the study
  * A NYHA classification of II controlled with treatment
  * Prior history of impaired cardiac function
* Participants may not have had a history of a stroke or transient ischemic attack within six months
* Participants should not have clinically significant peripheral vascular disease or vascular disease (including aortic aneurysm or aortic dissection)
* Participants may not have a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting cediranib
* Participants should not have any uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with untreated brain metastases, spinal cord compression, or evidence of symptomatic brain metastases or leptomeningeal disease as noted on computed tomography (CT) or magnetic resonance imaging (MRI) scans are ineligible; screening imaging to rule out brain metastases is not required for screening, but should be performed prior to study enrollment if clinically indicated; patients with treated brain metastases must demonstrate stable post-therapeutic imaging and resolution of any associated symptoms and must be stably off steroids with no symptoms for at least 6 months following therapy prior to starting study drug
* Participants may not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to cediranib or olaparib
* Participants receiving any medications or substances that are strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) or moderate inhibitors of CYP3A4 are ineligible; the study team should check a frequently-updated medical reference for a list of drugs to avoid or minimize use of; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product; dihydropyridine calcium-channel blockers are permitted for management of hypertension
* Pregnant women are excluded from this study because olaparib and cediranib have the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with olaparib and cediranib, breastfeeding should be discontinued if the mother is treated with cediranib and olaparib; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with cediranib or olaparib; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Participants should not have evidence of coagulopathy or bleeding diathesis; therapeutic anticoagulation for prior thromboembolic events is permitted
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment
  * Prophylactic use of bisphosphonates in patients without bone disease, except for the treatment of osteoporosis
  * Because the composition, PK, and metabolism of many herbal supplements are unknown, the concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, cannabis, St. John's wort, kava, ephedra [ma huang], ginkgo biloba, dehydroepiandrosterone [DHEA], yohimbe, saw palmetto, or ginseng)
  * Raloxifene is allowed for patients taking it for bone health
* Participants may not have any features suggestive of myelodysplastic syndrome (MDS) or acute myelogenous leukemia (AML) on peripheral blood smear or bone marrow biopsy, if clinically indicated

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2026-08-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce F Liu, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (20):
- United States (20):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 12 academic medical centers. The first participant was enrolled on May 23, 2016 and the last patient was enrolled on June 28, 2017.
Pre-assignment Details: A total of 70 participants enrolled to the study and received study intervention.
Groups:
- Cediranib/Olaparib in Platinum-Resistant Ovarian Cancer: Participants with platinum-resistant ovarian cancer received olaparib 200 mg orally twice daily and cediranib 30 mg orally once daily.
  Platinum-resistance is defined as disease progression within 6 months of platinum-based chemotherapy.
- Cediranib/Olaparib in Platinum-Sensitive Ovarian Cancer: Participants with platinum-sensitive ovarian cancer received olaparib 200 mg orally twice daily and cediranib 30 mg orally once daily.
  Platinum-sensitive disease is defined as cancer that has not progressed within 6 months of the last receipt of platinum-based chemotherapy.
Period: Overall Study
Arm/Group | Cediranib/Olaparib in Platinum-Resistant Ovarian Cancer | Cediranib/Olaparib in Platinum-Sensitive Ovarian Cancer
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cediranib/Olaparib in Platinum-Resistant Ovarian Cancer | Cediranib/Olaparib in Platinum-Sensitive Ovarian Cancer | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (9.47) | 59.4 (12.6) | 60.9 (11.1)
Age, Continuous [Median (Full Range); unit: years] | 62 [45 to 79] | 62 [33 to 76] | 62 [33 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 32 | 33 | 65
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 32 | 28 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70
BRCA Status [Count of Participants; unit: Participants]
  Wild Type | 22 | 12 | 34
  Mutation | 5 | 14 | 19
  Unknown | 8 | 9 | 17
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status
  0: Fully active, able to carry on all pre-disease performance without restriction
  1. Symptoms, but ambulatory. Restricted in physically strenuous activity but able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 28 | 24 | 52
    1 | 6 | 11 | 17
    2 | 1 | 0 | 1
Primary Site of Disease [Count of Participants; unit: Participants]
  Ovary | 33 | 29 | 62
  Fallopian Tube | 2 | 6 | 8
Number of Prior Lines [Count of Participants; unit: Participants] — Number of prior lines received of systemic chemotherapy.
  Participants
    1 | 14 | 14 | 28
    2 | 13 | 15 | 28
    3 | 6 | 5 | 11
    4 | 2 | 1 | 3
Platinum Status [Count of Participants; unit: Participants] — Platinum resistance is defined as disease that has progressed within 6 months of the last receipt of platinum-based chemotherapy. Platinum sensitivity is defined as cancer that has not progressed within 6 months of the last receipt of platinum-based chemotherapy.
  Participants
    Platinum Resistant | 35 | 0 | 35
    Platinum Sensitivity 6-12 Months | 0 | 24 | 24
    Platinum Sensitivity >12 Months | 0 | 11 | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) by HRR Status in Platinum-Sensitive Ovarian Cancer
Description: PFS determined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), where disease progression represents at least a 20% increase in the sum of diameters of target lesions, appearance of one or more new lesions, or unequivocal progression of existing non-target lesions.
  Homologous recombination repair (HRR) status was measured by the BROCA-HR assay. BROCA-HR is a targeted NGS platform including all known gynecologic cancer susceptibility genes and other DNA repair or related genes as well as a 3100 single nucleotide polymorphism panel to increase coverage for loss of heterozygosity (LOH) analysis. HRR status was associated as a pooled group against PFS using the Kaplan-Meier product-limit estimator with 95% confidence bands derived using Greenwood's formula.
Time Frame: Interval from start of treatment to documented disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death from any cause, whichever occurs first, assessed up to 32 months.
Population: Results are not reported for patients in the platinum-resistant ovarian cancer cohort as this primary objective pertained only to platinum-sensitive ovarian cancer.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- HRRmt: Genes included as homologous recombination repair mutant type (HRRmt): ATM, BARD1, BRCA1, BRCA2, BRIP1, CDK12 (somatic), NBN, PALB2, RAD51C, RAD51D
- HRRwt: homologous recombination repair wild type (HRRwt)
Arm/Group | HRRmt | HRRwt
Number analyzed (Participants) | 22 | 13
months | 16.79 [11.27 to 18.56] | 16.43 [9.4 to NA] — Not enough events to estimate upper confidence limit

2. Primary Outcome: Objective Response Rate (ORR) in Platinum-Resistant Ovarian Cancer
Description: Responses determined per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT or MRI, where Objective Response (OR) represents either a Complete Response (CR; disappearance of all target lesions) or a Partial Response (PR; at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum diameters); Objective Response (OR) = CR + PR.
Time Frame: Up to 32 months
Population: Results are not reported for patients in the platinum-sensitive ovarian cancer cohort as this primary objective pertained only to platinum-resistant ovarian cancer.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Platinum-Resistant Ovarian Cancer: Participants with platinum-resistant ovarian cancer received olaparib 200 mg orally twice daily and cediranib 30 mg orally once daily.
Arm/Group | Platinum-Resistant Ovarian Cancer
Number analyzed (Participants) | 35
percentage of participants | 22.86 [10.42 to 40.14]

3. Secondary Outcome: Biomarker Signature Development
Description: Will summarize the distribution of all candidate markers using descriptive statistics and non-parametric tests of their association with patient and disease characteristics. Biomarker profiles will be explored using unsupervised hierarchical clustering of all analytes and patients. The association of each candidate marker to progression-free survival will be evaluated by Cox proportional hazard models using a two-sided alpha = 0.05, while estimating the false discovery rate for any sets of identified markers by the Benjamini-Hochberg step-up procedure.
Time Frame: Up to 30 days post-treatment
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival
Description: Will be summarized using the Kaplan-Meier product-limit estimator with 95% confidence bands derived using Greenwood's formula.
Time Frame: Up to 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Genetic Alterations
Description: Will be detected by the BROCA-homologous recombination assay. Descriptive statistics will be used to summarize the genetic alterations detected by the BROCA-homologous recombination assay and Bioinformatics Pipeline. The prevalence of each genetic alteration will be reported overall, and within stratum defined by platinum-sensitive and platinum-resistant disease using binomial exact 95% confidence intervals. The primary analysis will associate BRCA mutations (germline or somatic) and other homologous recombination gene mutation (as a pooled group) with/against progression-free survival as a time-to-event endpoint, using Kaplan-Meier product-limit estimates and stratified logrank test using a two-sided alpha of 0.05.
Time Frame: Baseline
Reporting Status: Not Posted

6. Secondary Outcome: Change in Circulating Endothelial Cells/Circulating Endothelial Precursor Cells
Description: Will determine if there is an association between levels of circulating endothelial cells at baseline, or the change in circulating endothelial cells from baseline to day 3, and progression-free survival in patients receiving cediranib maleate/olaparib trial, and to determine if there are significant changes from baseline to day 3 in the levels of circulating endothelial cells. Will use a paired t-test. In addition, if the paired differences in values are not normally distributed (p < 0.05 by a Shapiro-Wilk test), then a Wilcoxon signed rank test will be used instead of a paired t-test.
Time Frame: Baseline to day 3
Reporting Status: Not Posted

7. Secondary Outcome: Prevalence of Genetic Alteration Using Whole Exome Sequencing
Description: The prevalence of each genetic alteration will be reported overall, and within platinum-sensitive and platinum-resistant cohorts using binomial exact 95% confidence intervals. Exploratory analyses will associate alterations of a single-gene against progression-free survival as a time-to-event endpoint, using Kaplan-Meier product-limit estimates and logrank test using a nominal two-sided alpha of 0.05.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout duration of therapy (up to 32 months).
Groups:
- Cediranib/Olaparib in Platinum-Sensitive Ovarian Cancer: Cediranib/Olaparib in Platinum-Sensitive Ovarian Cancer
  Participants with platinum-sensitive ovarian cancer received olaparib 200 mg orally twice daily and cediranib 30 mg orally once daily.
  Platinum-sensitive disease is defined as cancer that has not progressed within 6 months of the last receipt of platinum-based chemotherapy.
Arm/Group | Cediranib/Olaparib in Platinum-Sensitive Ovarian Cancer | Cediranib/Olaparib in Platinum-Resistant Ovarian Cancer
All-Cause Mortality (participants affected / at risk) | 9/35 | 12/35
Serious Adverse Events (participants affected / at risk) | 15/35 | 15/35
Other Adverse Events (participants affected / at risk) | 35/35 | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib/Olaparib in Platinum-Sensitive Ovarian Cancer (N=35) | Cediranib/Olaparib in Platinum-Resistant Ovarian Cancer (N=35)
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 5
Colitis (Gastrointestinal disorders) | 0 | 3
Colonic obstruction (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 0 | 2
GI Bleed (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
small intestinal obstruction (Gastrointestinal disorders) | 1 | 8
Vomiting (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
SIRS (Immune system disorders) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0
Concentration impairment (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cediranib/Olaparib in Platinum-Sensitive Ovarian Cancer (N=35) | Cediranib/Olaparib in Platinum-Resistant Ovarian Cancer (N=35)
Abdominal Distension (Cardiac disorders) | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 18 | 20
Activated Partial Thromboplastin Time Prolonged (Investigations) | 2 | 2
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 11 | 4
Alkaline Phosphatase Increased (Investigations) | 4 | 5
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 4
Amnesia (Nervous system disorders) | 1 | 0
Amotivation (General disorders) | 1 | 0
Anal Hemorrhage (Gastrointestinal disorders) | 1 | 1
Anemia (Blood and lymphatic system disorders) | 8 | 7
Anorexia (Metabolism and nutrition disorders) | 21 | 11
Anxiety (Psychiatric disorders) | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 4
Ascites (Gastrointestinal disorders) | 1 | 2
Aspartate Aminotransferase Increased (Investigations) | 8 | 7
Athralgia (General disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 6
Bloating (Gastrointestinal disorders) | 6 | 6
Blood Bilirubin Increased (Investigations) | 1 | 0
Blurred Vision (Eye disorders) | 3 | 2
Brain Fog (General disorders) | 3 | 0
Bruising (Injury, poisoning and procedural complications) | 4 | 2
Burning Eyes (Eye disorders) | 4 | 1
Cellulitis (Infections and infestations) | 1 | 0
Chest Pain - Cardiac (Cardiac disorders) | 1 | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Chills (General disorders) | 2 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 2 | 0
Cognitive Disturbance (Nervous system disorders) | 2 | 1
Cold Symptoms (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Colonic Fistula (Gastrointestinal disorders) | 1 | 0
Concentration Impairment (Nervous system disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 16
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Creatinine Increased (Investigations) | 6 | 2
Critical High Lactic Acid (Investigations) | 1 | 0
Cystitis Noninfective (Renal and urinary disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 5 | 4
Depression (Psychiatric disorders) | 4 | 3
Diarrhea (Gastrointestinal disorders) | 34 | 30
Dizziness (Nervous system disorders) | 7 | 6
Dry Mouth (Gastrointestinal disorders) | 6 | 3
Dry Nipples (Skin and subcutaneous tissue disorders) | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 0
Dysesthesia (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 7 | 7
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 10
Ear Pain (Ear and labyrinth disorders) | 1 | 1
Edema Limbs (General disorders) | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema (Eye disorders) | 1 | 0
Eye Hemorrhage (Eye disorders) | 1 | 0
Face Numbness (Nervous system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Fatigue (General disorders) | 31 | 26
Fever (General disorders) | 3 | 1
Flatulence (Gastrointestinal disorders) | 4 | 1
Flu Like Symptoms (General disorders) | 2 | 2
Flushing (Vascular disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 5
Gastroparesis (Gastrointestinal disorders) | 1 | 0
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 3
GI Bleed (Gastrointestinal disorders) | 1 | 0
Gum Infection (Infections and infestations) | 1 | 0
Head Cold (General disorders) | 1 | 0
Headache (Nervous system disorders) | 13 | 12
Hematuria (Renal and urinary disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 7 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 4 | 3
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 2 | 0
Hypertension (Vascular disorders) | 24 | 23
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 2
Hyponatremia (Metabolism and nutrition disorders) | 5 | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 3 | 2
Hypotension (Vascular disorders) | 4 | 5
Hypothyroidism (Endocrine disorders) | 16 | 9
Increased Phosphorus (Blood and lymphatic system disorders) | 1 | 0
Increased TSH (Investigations) | 2 | 1
Indigestion (General disorders) | 1 | 0
Insect Bites (Skin and subcutaneous tissue disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 2
L Rotator Cuff Tear (General disorders) | 3 | 0
L Rotator Cuff Tear (Musculoskeletal and connective tissue disorders) | 3 | 0
Laryngeal Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Left Eye Erythema (Eye disorders) | 1 | 0
Left Face Numbness (Nervous system disorders) | 1 | 0
Left Rotator Cuff Tear (Musculoskeletal and connective tissue disorders) | 1 | 0
Lightheadedness (General disorders) | 1 | 0
Lips/Tongue Numbness (Nervous system disorders) | 3 | 0
Lower Extremity Swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung Infection (Infections and infestations) | 2 | 0
Lymphocyte Count Decreased (Investigations) | 6 | 4
Malaise (General disorders) | 1 | 1
Memory Impairment (Nervous system disorders) | 1 | 2
Mucosal Infection (Infections and infestations) | 2 | 0
Mucositis Oral (Gastrointestinal disorders) | 13 | 6
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 1
Nail Discoloration (Skin and subcutaneous tissue disorders) | 1 | 0
Nail Infection (Infections and infestations) | 1 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 30 | 22
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Neutrophil Count Decreased (Investigations) | 8 | 8
Non-Cardiac Chest Pain (General disorders) | 5 | 1
Numbness Left Side of Face (Nervous system disorders) | 2 | 0
Oral Pain (Gastrointestinal disorders) | 2 | 1
Pain (General disorders) | 5 | 9
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 9 | 7
Palmar-Plantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 6 | 6
Palpitations (Cardiac disorders) | 1 | 1
Paresthesia (Nervous system disorders) | 3 | 0
Pelvic Pain (Reproductive system and breast disorders) | 1 | 3
Peripheral Motor Neuropathy (Nervous system disorders) | 1 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 7 | 1
Platelet Count Decreased (Investigations) | 6 | 8
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Proteinuria (Renal and urinary disorders) | 5 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Acneiform (Skin and subcutaneous tissue disorders) | 2 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 2
Rectal Hemorrhage (Gastrointestinal disorders) | 2 | 1
Rectal Pain (Gastrointestinal disorders) | 1 | 0
Renal Calculi (Renal and urinary disorders) | 1 | 0
Right Eye Hemorrhage (Eye disorders) | 4 | 0
Rotator Cuff (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator Cuff Tear (Musculoskeletal and connective tissue disorders) | 1 | 0
Salivary Duct Inflammation (Gastrointestinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Sinus Bradycardia (Cardiac disorders) | 1 | 1
Sinus Pain (Nervous system disorders) | 1 | 0
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Sinusitis (Infections and infestations) | 4 | 0
SIRS (Immune system disorders) | 1 | 0
Skin Infection (Infections and infestations) | 1 | 0
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 7
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Stomach Pain (Gastrointestinal disorders) | 2 | 0
Thromboembolic Event (Vascular disorders) | 2 | 1
Thrombotic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 0
Thrush (Infections and infestations) | 1 | 1
Tongue Discoloration (Gastrointestinal disorders) | 1 | 0
Tongue Discoloration (General disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Total Protein Decreased (Investigations) | 1 | 0
TSH Increased (Investigations) | 2 | 0
Upper Respiratory Infection (Infections and infestations) | 3 | 3
Urinary Burning (Renal and urinary disorders) | 1 | 0
Urinary Frequency (Renal and urinary disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 8 | 5
Urinary Tract Pain (Renal and urinary disorders) | 1 | 1
Urinary Urgency (Renal and urinary disorders) | 1 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal Dryness (Reproductive system and breast disorders) | 1 | 1
Vaginal Hemorrhage (Reproductive system and breast disorders) | 2 | 0
Vaginal Infection (Infections and infestations) | 1 | 0
Vaginal Pain (Reproductive system and breast disorders) | 1 | 0
Voice Alteration (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 18 | 19
Weight Loss (Investigations) | 4 | 5
White Blood Cell Decreased (Investigations) | 7 | 5
Yeast Infection (Infections and infestations) | 1 | 0
Bronchial Infection (Infections and infestations) | 0 | 1
Burning Eyes (Injury, poisoning and procedural complications) | 4 | 1
Cholesterol High (Investigations) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 4
Colonic Obstruction (Gastrointestinal disorders) | 0 | 2
Colorful Blotches in Vision (Eye disorders) | 0 | 1
Early Satiety (Gastrointestinal disorders) | 0 | 3
Elevated Thyroid (Investigations) | 0 | 2
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Floaters (Eye disorders) | 0 | 1
Floaters and Changes in Depth Perception (Eye disorders) | 0 | 1
Flu (Infections and infestations) | 0 | 1
Gait Disturbance (General disorders) | 0 | 1
Hemoglobin Increased (Investigations) | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hot Flashes (Vascular disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1
Increased TSH (Endocrine disorders) | 2 | 1
Lipase Increased (Investigations) | 0 | 1
Localized Edema (General disorders) | 0 | 1
Lower Respiratory Infection (Infections and infestations) | 0 | 1
Muscle Aching (Musculoskeletal and connective tissue disorders) | 0 | 2
Periorbital Edema (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rotator Cuff Injury (Musculoskeletal and connective tissue disorders) | 0 | 2
Seizure (Nervous system disorders) | 0 | 1
Split Tongue (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/65/NCT02345265/Prot_SAP_000.pdf